CLINICAL TRIAL: NCT03749993
Title: Evaluation of a MRI-based Prostate Cancer Screening Program
Acronym: VISIONING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VISIONING1
Record Dates: First submitted 2018-09-24; First posted 2018-11-21 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Arm (Other): Screening
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Use of bpMRI for opportunistic prostate cancer screening.

SUMMARY:
The purpose of this study is to evaluate the effort and resources (incl. costs) required to detect 20 clinically relevant prostate cancer (PCA) in a screening program based on bpMRI of the prostate.

DETAILED DESCRIPTION:
Informed men at risk for prostate cancer will be included into the study to undergo prostate cancer screening. According to European guidelines we will include men > 50 years of age and men >45 years of age and a family history of PCA as well as African-Americans >45 years of age. In this study, bpMRI will be used for opportunistic prostate cancer screening.

The indication for prostate biopsy is based solely on the results of bpMRI. In case of detection of lesions suspicious for prostate cancer ( PIRADS 3), targeted MRI-TRUS fusion biopsy with 3 biopsies per lesion will be performed. In case no lesions suspicious for PCA ( PIRADS 3) are detected, SB will performed if PSA exceeds 10ng/ml and/or DRE is suspicious for PCA.

ELIGIBILITY:
Inclusion Criteria:

* well-informed men with the wish for prostate cancer screening
* prostate biopsy naïve
* life expectancy > 10 years
* men > 50 years of age
* men > 45 years of age with a family history of prostate cancer
* African-Americans > 45 years of age

Exclusion Criteria:

* prostate biopsy performed prior to study
* life expectancy < 10 years
* acute urinary tract infection
* NIH-CPSI score 19 (leads to initiation of urologic diagnostics and treatment)
* IPSS score 20 (leads to initiation of urologic diagnostics and treatment)

Contraindications for MRI:

* Heart pacemaker
* Artificial heart valves (some types are eligible)
* Cochlea implant
* ICD
* Metallic foreign bodies/devices/implants (neuro-stimulator, pain or insulin pump, etc.)
* Severe claustrophobia

Ages: 46 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Informed men at risk for prostate cancer will be included into the study to undergo prostate cancer screening.
Enrollment: 241 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Total costs of the MRI based prostate cancer screening | 24 months
  Total costs of the program

SECONDARY OUTCOMES:
Comparison of costs of classical screening based on PSA and DRE | 24 months
  Total costs per patient
number of patients undergoing active surveillance | 24 months
  Number of follow-up interventions
number of patients undergoing radical cystoprostatectomy | 24 months
  Number of follow-up interventions
number of patients undergoing radiotherapy | 24 months
  Number of follow-up interventions
number of patients undergoing androgen deprivation therapy | 24 months
  Number of follow-up interventions
number of patients undergoing chemotherapy | 24 months
  Number of follow-up interventions
Quality of Life (Qol) | 24 months
  Qol Questionnaire (SF- 36) score (0-100), 0 means best, 100 worst case
Distress Thermometer Assessment | 24 months
  "Distress Thermometer" score (0-10)
AI Evaluation | 24 months
  Evaluation of algorithms (AI) for CAD MRI based PCA diagnostic
Number of patients | 24 months
  Number of patients needed to screen
Number of consultations | 24 months
  Number of total consultations

CONTACTS AND LOCATIONS:
Overall Officials: Cyrill Rentsch, MD PHD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinic of Urology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No